CLINICAL TRIAL: NCT02795065
Title: Bemiparin Versus Enoxaparin in the Prevention of Venous Thromboembolism Among ICU Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamed Sayed Mohamed Abbas (Other)
Responsible Party: Sponsor-Investigator, Mohamed Sayed Mohamed Abbas, Doctor, Al Mouwasat Hospital
Organization: Al Mouwasat Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSAT-4
Record Dates: First submitted 2016-06-06; First posted 2016-06-09 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Enoxaparin; bemiparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enoxaparin 40 mg subcutaneous once daily (Active Comparator)
  Interventions: Drug: Enoxaparin
- Bemiparin 3500 IU subcutaneous once daily (Experimental)
  Interventions: Drug: Bemiparin

INTERVENTIONS:
Drug: Enoxaparin — Use of enoxaparin 40 mg subcutaneous once daily in high risk intensive care patients as a prophylaxis against venous thromboembolism
  Arms: Enoxaparin 40 mg subcutaneous once daily
Drug: Bemiparin — Use of bemiparin 3500 IU subcutaneous once daily in high risk intensive care patients as a prophylaxis against venous thromboembolism
  Arms: Bemiparin 3500 IU subcutaneous once daily

SUMMARY:
The purpose of this study is to compare two types of low-molecular-weight heparin, enoxaparin and bemiparin, as regards their efficacy and safety in venous thromboembolism prevention among intensive care unit patients.

DETAILED DESCRIPTION:
A prospective randomized trial to compare thromboprophylaxis using bemiparin and enoxaparin in critically ill patients in ICU. The study included one hundred bedridden patients in intensive care unit who are at high risk for developing venous thromboembolism and require long term anticoagulation

Patients were divided into two groups each one consists of 50 patients. One group received bemiparin 3500 IU subcutaneous once daily and the other group received enoxaparin 40 mg subcutaneous once daily as a prophylaxis against thromboembolism.

Patients were followed up for 60 days for the development of deep venous thrombosis, pulmonary embolism and complications related to the injected anticoagulant.

ELIGIBILITY:
Inclusion Criteria:

* Sepsis , stroke , major burn , respiratory failure , traumatic brain injury , malignancy and post arrest who are intubated and mechanically ventilated on continuous IV sedation

Exclusion Criteria:

* Hypersensitivity to low molecular weight heparins , hypercoagulability , congenital or acquired bleeding disorder, prolongation of activated partial thromboplastin time or prothrombin time by 20% compared to normal values; thrombocytopenia (platelet count <100,000/mm3); macroscopic hematuria; uncontrolled hypertension [systolic blood pressure >200 mmHg; diastolic blood pressure >100 mmHg]; impaired kidney function: serum creatinine > 2.0 mg/ dL and bleeding gastrointestinal ulcer.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Development of deep venous thrombosis | Within 2 years
  Deep venous thrombosis was detected using bilateral lower limb venous duplex done twice weekly over the period of 60 days or if patient had clinical symptoms of deep venous thrombosis during hospitalization. Best evaluation of Different lower extremities veins is obtained by using different ultrasound techniques. Proximal deep veins, specifically the common femoral, femoral, and popliteal veins are usually examined using compression ultrasound whereas a combination of duplex ultrasound and color Doppler imaging is more often used to interrogate the calf and iliac veins
Development of pulmonary embolism | Within 2 years
  Pulmonary embolism was detected clinically by hypotension, tachycardia, hypoxemia, and decreased end-tidal carbondioxide and confirmed radiologically by CT pulmonary angiography if there was arterial occlusion with failure to enhance the entire lumen due to a large filling defect , a partial filling defect surrounded by contrast material or a peripheral intraluminal filling defect that forms acute angles with the arterial wall
Complications related to the injected anticoagulant | Within 2 years
  Patient were followed up daily for complications related to the injected anticoagulant including any ecchymosis or hematomas developed at the site of anticoagulant injection , the presence of major bleeding defined as decrease in hemoglobin levels by 2 gm/L or more or requiring transfusion of 2 or more units of packed red cells or whole blood, the presence of minor bleeding defined as any bleeding other than major bleeding events , drop in the platelet count and the presence of allergic skin reactions or urticaria, If any of these complications was observed , the anticoagulant was immediately discontinued.

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Navarro-Quilis A, Castellet E, Rocha E, Paz-Jimenez J, Planes A; Bemiparin Study Group in Knee Arthroplasty. Efficacy and safety of bemiparin compared with enoxaparin in the prevention of venous thromboembolism after total knee arthroplasty: a randomized, double-blind clinical trial. J Thromb Haemost. 2003 Mar;1(3):425-32. doi: 10.1046/j.1538-7836.2003.00142.x. PMID 12871445
- [Derived] Abbas MS. Bemiparin versus Enoxaparin in the Prevention of Venous Thromboembolism among Intensive Care Unit Patients. Indian J Crit Care Med. 2017 Jul;21(7):419-423. doi: 10.4103/ijccm.IJCCM_23_17. PMID 28808360